CLINICAL TRIAL: NCT01993888
Title: A Phase III Randomized, Controlled, Superiority Study Evaluating EVARREST® Fibrin Sealant Patch Versus Standard of Care Treatment in Controlling Parenchymal Bleeding During Hepatic Surgery
Brief Title: The EVARREST® Fibrin Sealant Patch Liver Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOS-13-005; 2013-002535-24 (EudraCT Number)
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-04

CONDITIONS: Hemorrhage
Keywords: Hepatobiliary Surgery
MeSH Terms: conditions — Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVARREST® Fibrin Sealant Patch (Experimental): EVARREST® Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts - a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Interventions: Biological: EVARREST® Fibrin Sealant Patch
- Standard of Care (SoC) (Other): SoC is a composite of techniques/methods typically used by the surgeon to control bleeding after conventional methods (i.e. suture, ligation, cautery) are ineffective or impractical. For this study, SoC will be initiated with continuous firm manual compression with or without gauze or sponge and with or without a topical absorbable hemostat (example SURGICEL).
  Interventions: Other: Standard of Care (SoC)

INTERVENTIONS:
Biological: EVARREST® Fibrin Sealant Patch
  Arms: EVARREST® Fibrin Sealant Patch
Other: Standard of Care (SoC)
  Arms: Standard of Care (SoC)

SUMMARY:
To evaluate the safety and hemostatic effectiveness of EVARREST® Fibrin Sealant Patch (EVARREST) versus standard of care treatment (SoC) in controlling parenchymal bleeding during hepatic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age, requiring elective or urgent, open hepatic surgery.
* Presence of an appropriate bleeding hepatic parenchymal Target Bleeding Site (TBS) as identified intra-operatively by the surgeon
* Subjects or legally authorized representatives must be willing to participate in the study, and provide written informed consent. (Note: This criteria does allow for hospital translators to be used where approved by Ethics Committees/Institutional Review Boards)

Exclusion Criteria:

* Subjects with any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure;
* TBS is from large defects in arteries or veins where the injured vascular wall requires repair with maintenance of vessel patency and which would result in persistent exposure of EVARREST® to blood flow and pressure during healing and absorption of the product;
* TBS with major arterial bleeding requiring suture or mechanical ligation;
* Subjects admitted for trauma surgery;
* Subject is a transplant patient for fulminant hepatic failure
* Subject with TBS within an actively infected field;
* Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine;
* Subjects with known intolerance to blood products or to one of the components of the study product or is unwilling to receive blood products;
* Subjects who are known, current alcohol and / or drug abusers;
* Subjects who have participated in another investigational medical device or investigational drug trial within 30 days of surgery or are expected to participate in another medical device or investigational drug trial during the course of the study;
* Female subjects who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, Study Director — Ethicon, Inc.
Locations (17):
- United States (10):
  - Clinical Investigation Site #13, Birmingham, Alabama
  - Clinical Investigation Site #10, Augusta, Georgia
  - Clinical Investigation Site #16, Chicago, Illinois
  - Clinical Investigation Site #12, Chicago, Illinois
  - Clinical Investigation Site #15, New Orleans, Louisiana
  - Clinical Investigation Site #9, St Louis, Missouri
  - Clinical Investigation Site #11, New York, New York
  - Clinical Investigation Site #14, New York, New York
  - Clinical Investigation Site #8, Philadelphia, Pennsylvania
  - Clinical Investigation Site #17, Pittsburgh, Pennsylvania
- Australia (2):
  - Clinical Investigation Site #3, Melbourne
  - Clinical Investigation Site #2, Woodville South
- Clinical Investigation Site #1, Auckland, New Zealand
- United Kingdom (4):
  - Clinical Investigation Site #6, Birmingham
  - Clinical Investigation Site #7, Cambridge
  - Clinical Investigation Site #4, Edinburgh
  - Clinical Investigation Site #5, Leeds

REFERENCES:
- [Result] Koea JB, Batiller J, Aguirre N, Shen J, Kocharian R, Bochicchio G, Garden OJ. A multicentre, prospective, randomized, controlled trial comparing EVARREST fibrin sealant patch to standard of care in controlling bleeding following elective hepatectomy: anatomic versus non-anatomic resection. HPB (Oxford). 2016 Mar;18(3):221-8. doi: 10.1016/j.hpb.2015.12.006. Epub 2016 Feb 1. PMID 27017161
- [Derived] Corral M, Ferko N, Hollmann S, Hogan A, Jamous N, Batiller J, Shen J. Clinician reported ease of use for a novel fibrin sealant patch for hemostasis: results from four randomized controlled trials. Curr Med Res Opin. 2016;32(2):367-75. doi: 10.1185/03007995.2015.1128405. Epub 2015 Dec 21. PMID 26636489

RESULTS

PARTICIPANT FLOW:
Groups:
- EVARREST Fibrin Sealant Patch: EVARREST™ Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts - a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  EVARREST™ Fibrin Sealant Patch
- Standard of Care (SoC): SoC is a composite of techniques/methods typically used by the surgeon to control bleeding after conventional methods (i.e. suture, ligation, cautery) are ineffective or impractical. For this study, SoC will be initiated with continuous firm manual compression with or without gauze or sponge and with or without a topical absorbable hemostat (example SURGICEL).
  Standard of Care (SoC)
Period: Overall Study
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Started | 50 | 52
Completed | 48 | 49
Not Completed | 2 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC) | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 24 | 24 | 48
Age, Continuous [Mean (Full Range); unit: years] | 61.3 [23 to 81] | 63.2 [36 to 85] | 62.2 [23 to 85]
Age, Continuous [Median (Standard Deviation); unit: years] | 64 (14.5) | 63 (10.9) | 63 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 30 | 32 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 43 | 44 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  New Zealand | 6 | 7 | 13
  United States | 18 | 18 | 36
  United Kingdom | 15 | 15 | 30
  Australia | 11 | 12 | 23
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 28 (5.6) | 28.1 (5.9) | 28 (5.7)
BMI (kg/m2) [Median (Full Range); unit: kg/m^2] | 27.5 [17.5 to 43.3] | 26.8 [15.2 to 42.5] | 27.4 [15.2 to 43.3]
BMI (Grouped) [Number; unit: participants]
  Underweight | 2 | 2 | 4
  Normal | 13 | 14 | 27
  Overweight | 19 | 16 | 35
  Obese | 14 | 18 | 32
  Morbidly Obese | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 4-minutes Following Randomization
Description: Proportion of subjects achieving hemostasis at the TBS at 4-minutes following randomization and with no re-bleeding requiring treatment at the TBS any time prior to initiation of wound closure. Hemostasis is defined as no detectable bleeding at the TBS.
Time Frame: Intraoperative, 4 minutes following randomization
Population: The primary endpoint analysis was based on the Intent to Treat (ITT) analysis set.
Measure: Number; unit: participants with hemostatic success
Groups:
- EVARREST™ Fibrin Sealant Patch: EVARREST™ Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts - a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
Arm/Group | EVARREST™ Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 50 | 52
participants with hemostatic success | 48 | 24
Statistical Analysis 1: Comparison: EVARREST™ Fibrin Sealant Patch vs Standard of Care (SoC); Test type: Superiority or Other; p < .0001, Chi-squared

2. Secondary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 10-minutes Following Randomization
Description: Proportion of subjects achieving hemostatic success at 10 minutes following randomization and no further bleeding requiring treatment prior to initiation of wound closure.
Time Frame: Intraoperative, 10 minutes following randomization
Population: The proportion of subjects achieving hemostatic success at 10 minutes following randomization was evaluated as a secondary endpoint using the logistic model with treatment and site/institution included in the model.
Measure: Number; unit: participants with hemostatic success
Arm/Group | EVARREST™ Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 50 | 52
participants with hemostatic success | 49 | 42

3. Secondary Outcome: Absolute Time to Hemostasis
Description: The absolute time to achieve hemostasis at or after 4 minutes from randomization.
Time Frame: Intraoperative, an average of 4.2 minutes following randomization
Population: Time to hemostasis (TTH), defined as the absolute time to achieve hemostasis at or after 4 minutes from randomization was evaluated as a secondary endpoint. In one subject in the SoC group, manual compression was not maintained until the 4-minute endpoint, but was released early and a suture was applied, at which point the subject was hemostatic.
Measure: Median (Full Range); unit: minutes
Arm/Group | EVARREST™ Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 50 | 51
minutes | 4.0 [4.0 to 15.9] | 4.7 [1.7 to 33.0]

4. Secondary Outcome: Incidence of Re-bleeding Events From the TBS During the Study Follow-up
Time Frame: Up to 60-days following surgery
Measure: Number; unit: participants
Arm/Group | EVARREST™ Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 50 | 52
participants
  Continuous bleeding | 1 | 24
  Re-bleeding | 0 | 3
  Durability of hemostasis | 1 | 1
  Application error | 0 | 1

5. Secondary Outcome: Incidence of Adverse Events (AEs)
Time Frame: Up to 60-days following surgery
Measure: Number; unit: participants
Arm/Group | EVARREST™ Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 50 | 52
participants
  Participants experienced at least one AE | 45 | 50
  Participants experienced at least one SAE | 12 | 16
  Participants experienced at least one Severe AE | 8 | 6

6. Secondary Outcome: Incidence of Adverse Events That Were Potentially Related to Thrombotic Events
Description: Number of participants with adverse events that were potentially related to thrombic events
Time Frame: Up to 60-days following surgery
Measure: Number; unit: participants
Arm/Group | EVARREST™ Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 50 | 52
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of randomization until 60 days following the study procedure.
Groups:
- EVARREST Fibrin Sealant Patch: EVARREST™ Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts - a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Serious Adverse Events (participants affected / at risk) | 12/50 | 16/52
Other Adverse Events (participants affected / at risk) | 45/50 | 50/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVARREST Fibrin Sealant Patch (N=50) | Standard of Care (SoC) (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Localized Intraabdominal Fluid Collection (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Haematoma Infection (Infections and infestations) | 2 | 0
Liver Abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 0 | 2
Subdiaphragmatic Abscess (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Chemical Peritonitis (Injury, poisoning and procedural complications) | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1
Post-procedural Bile Leak (Injury, poisoning and procedural complications) | 2 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 | 1
Wound Decomposition (Injury, poisoning and procedural complications) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 2
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVARREST Fibrin Sealant Patch (N=50) | Standard of Care (SoC) (N=52)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Leukocytosis (Blood and lymphatic system disorders) | 3 | 2
Atrial Fibrillation (Cardiac disorders) | 2 | 4
Bradycardia (Cardiac disorders) | 1 | 3
Tachycardia (Cardiac disorders) | 4 | 11
Abdominal Distension (Gastrointestinal disorders) | 2 | 3
Abdominal Pain (Gastrointestinal disorders) | 5 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Acites (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 14 | 22
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Nausea (Gastrointestinal disorders) | 25 | 23
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 13 | 14
Oedema (General disorders) | 4 | 1
Odema Peripheral (General disorders) | 5 | 3
Pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 13 | 11
Pneumonia (Infections and infestations) | 3 | 3
Urinary Tract Infection (Infections and infestations) | 2 | 5
Wound Infection (Infections and infestations) | 1 | 3
Post-procedural Bile Leak (Injury, poisoning and procedural complications) | 2 | 3
Postoperative Ileus (Injury, poisoning and procedural complications) | 3 | 4
Procedural Pain (Injury, poisoning and procedural complications) | 5 | 10
Wound Secretion (Injury, poisoning and procedural complications) | 3 | 4
Blood Lactic Acid Increased (Investigations) | 4 | 6
International Normalized Ratio Increased (Investigations) | 4 | 2
Urine Output Decreased (Investigations) | 4 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 11
Malnutrition (Metabolism and nutrition disorders) | 3 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Dizziness (Nervous system disorders) | 6 | 6
Lethargy (Nervous system disorders) | 1 | 3
Confusional State (Psychiatric disorders) | 3 | 6
Hallucination (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 5 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 7
Hypertension (Vascular disorders) | 6 | 5
Hypotension (Vascular disorders) | 14 | 18

LIMITATIONS AND CAVEATS:
* The study could not be blinded due to difference in groups
* The efficacy was limited to one bleeding site to minimize the variability in assessing the primary endpoint
* The sample may not be sufficient to detect a difference in clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less